CLINICAL TRIAL: NCT02820597
Title: Clinical Evaluation of Cryotherapy in the Nasal Passageway Using the ClariFix Device
Brief Title: ClariFix Cryoablation Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arrinex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2014-02
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): Cryoablation with the ClariFix device
  Interventions: Device: ClariFix device

INTERVENTIONS:
Device: ClariFix device

SUMMARY:
This is a single-arm pilot study designed to evaluate the feasibility of cryoablation in the nasal passageway, using the ClariFix device, to reduce the symptoms of chronic rhinitis.

DETAILED DESCRIPTION:
This is a small, prospective, multicenter, single-arm, self-controlled interventional feasibility study to evaluation cryoablation in the nasal passage as a treatment for chronic rhinitis. The ClariFix device is FDA-cleared device with the intended use for the destruction of unwanted tissue during surgical procedures, including in adults with chronic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is >21 years of age
2. Subject has had moderate to severe symptoms of rhinorrhea and/or nasal congestion for >3 months (rTNSS rating of 2 or 3)
3. Subject has signed IRB-approved informed consent form

Exclusion Criteria:

1. Subject has clinically significant anatomic obstructions that limit access to the posterior nose including severe septal deviation, nasal polyps, and sinonasal tumor
2. Subject has a septal perforation
3. Subject has had prior sinus or nasal surgery that significantly alters the anatomy of the posterior nose
4. Subject has had prior head or neck irradiation
5. Subject has active or chronic nasal or sinus infection
6. Subject has active coagulation disorder or patient is receiving anti-coagulants which cannot be safely stopped for 2 weeks
7. Subject has a history of dry nose symptoms
8. Subject is pregnant or lactating
9. Subject is participating in another clinical research study
10. Subject has an allergy or intolerance to anesthetic agent
11. Subject is an active smoker or has been a smoker within the last 6 months
12. Any physical condition that in the investigator's opinion would prevent adequate study participation or pose increased risk

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2016-02-05 (Actual); Study Completion 2016-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Johnson, MD, Principal Investigator — San Francisco Otolaryngology Medical Group

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hwang PH, Lin B, Weiss R, Atkins J, Johnson J. Cryosurgical posterior nasal tissue ablation for the treatment of rhinitis. Int Forum Allergy Rhinol. 2017 Oct;7(10):952-956. doi: 10.1002/alr.21991. Epub 2017 Aug 11. PMID 28799727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 participants were enrolled and treated with bilateral cryotherapy of the nasal passage (54 treatments).
Period: Overall Study
Arm/Group | Intervention
Started | 27
1-day Post Treatment | 27
7-day Post Treatment | 27
30-day Post Treatment | 27
90-day Post Treatment | 24 (2 participants missed the 90-day visit, 1 participant was lost to follow-up.)
180-day Post Treatment (Initially, study was complete upon 90 days follow-up, the 180-day visit was added later.) | 21 (3 participants missed the 180-day visit, 3 participants were lost to follow-up.)
Completed (Initially, study was complete upon 90 days follow-up, the 365-day visit was added later.) | 15 (12 participants were lost to follow-up.)
Not Completed | 12
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Treatment with the ClariFix Device
  ClariFix Device
Arm/Group | Intervention
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: Years] | 53.29 [27 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Device- and/or Procedure-related Serious Adverse Events
Description: Number of participants with device- and/or procedure-related serious adverse events reported over the initial study follow-up period.
Time Frame: Baseline through 365 days post treatment
Population: A total of 27 subjects were enrolled and received bilateral cryosurgery with the ClariFix device (n=54 treatments).
Measure: Number; unit: participants
Arm/Group | Intervention
Number analyzed (Participants) | 27
participants | 0

2. Primary Outcome: Change in Rhinitis Symptom Severity (rTNSS)
Description: Change from baseline in participant-reported symptom severity based on the rTNSS (Reflective Total Nasal Symptom Score). The rTNSS is the sum of 4 individual subject-assessed symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, each evaluated using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe. The rTNSS has a possible score range of 0-12. The reflective scores are based on the participant's evaluation of symptom severity over the preceding 12 hours.
Time Frame: Baseline through 365 days post treatment
Population: All participants with follow-up at the indicated visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 27
score on a scale
  7 Days post treatment | -1.9 (0.6)
  30 Days post treatment | -3.6 (0.6)
  90 Days post treatment: number analyzed (Participants) | 24
  90 Days post treatment | -3.3 (0.6)
  180 Days post treatment: number analyzed (Participants) | 21
  180 Days post treatment | -4.0 (0.5)
  365 Days post treatment: number analyzed (Participants) | 15
  365 Days post treatment | -4.5 (0.3)
Statistical Analysis 1: Comparison: Intervention; Null hypothesis is that the within-participant change from baseline in rTNSS is 0; Test type: Superiority; p < 0.001, t-test, 2 sided; Paired t-tests on the mean change from baseline. No adjustments were made for multiple comparisons

3. Primary Outcome: Change in Rhinitis Symptoms (VAS)
Description: Change from baseline in rhinitis symptoms measured on a participant-reported visual analog scale (VAS). Symptoms of rhinorrhea, nasal breathing, facial pain/pressure, and sense of smell were rated from 0 (no symptoms) to 10 (severe/extremely bothersome symptoms) assessed over the 12 hours preceding the visit. An average of the 4 individual scores was used as the total VAS score with a range of 0 to 10.
Time Frame: Baseline through 365 days post treatment
Population: All treated participants with follow-up at the indicated visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 27
score on a scale
  7 Days post treatment | -2.1 (0.5)
  30 Days post treatment | -3.8 (0.5)
  90 Days post treatment: number analyzed (Participants) | 24
  90 Days post treatment | -4.1 (0.6)
  180 Days post treatment: number analyzed (Participants) | 21
  180 Days post treatment | -2.9 (0.7)
  365 Days post treatment: number analyzed (Participants) | 15
  365 Days post treatment | -5.6 (1.1)
Statistical Analysis 1: Comparison: Intervention; Null hypothesis is that the within-participant change from baseline in rhinitis symptoms VAS is 0; Test type: Superiority; p < 0.001, t-test, 2 sided — Paired t-tests on the mean change from baseline. No adjustments were made for multiple comparisons

4. Secondary Outcome: Ease of Use
Description: Physician evaluation of ClariFix ease of use. After each participant's treatment, the physician was asked to rate the ClariFix on ease of use. Options were easy, moderately easy, moderately difficult, or difficult.
Time Frame: Immediately post treatment
Population: Physician evaluation of ease of use after each ClariFix procedure.
Measure: Count of Units; unit: Procedures
Units Other Than Participants: Procedures
Arm/Group | Intervention
Number analyzed (Participants) | 27
Number analyzed (Procedures) | 27
Procedures
  Easy | 14
  Moderately easy | 10
  Moderately difficult | 3
  Difficult | 0

5. Secondary Outcome: Device- and/or Procedure-related Adverse Events
Description: All adverse events evaluated as possibly, probably, or definitely related to the ClariFix device and/or procedure.
Time Frame: Baseline through 90 days post treatment
Population: All treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 27
Participants | 1

ADVERSE EVENTS:
Time Frame: 1 Year
Description: Adverse events were systematically reported at each follow-up visit.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 19/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=27)
Ear blockage (General disorders) | 12 (12)
Nasal Dryness (General disorders) | 7 (7)
Epitaxsis (General disorders) | 1 (1) — Moderate nosebleed

LIMITATIONS AND CAVEATS:
This is a feasibility study based on a small population of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes